CLINICAL TRIAL: NCT02284919
Title: Imaging of In Vivo Sigma-2 Receptor Expression With [18F]ISO-1 Positron Emission Tomography (PET/CT) in Primary Breast Cancer
Brief Title: [18F]ISO-1 Positron Emission Tomography (PET/CT) in Primary Breast Cancer
Acronym: ISO-1Primary
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 820737; NCT02762110 (obsolete NCT alias)
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ISO-1 PET/CT (Experimental): All subjects will receive an [18F]ISO-1 PET/CT scan
  Interventions: Drug: [18F]ISO-1

INTERVENTIONS:
Drug: [18F]ISO-1 — [18F]ISO-1 PET/CT scan
  Other Names: N-(4-(6,7-dimethoxy-3,-4-dihydroisoquinolin-2(1H)-yl)butyl)-2-(2-[18F]-fluoroethoxy)-5- Methylbenzamide ([18F]ISO-1)

SUMMARY:
In this study, positron emission tomography (PET/CT) imaging will be used to evaluate sigma-2 (σ2) receptor activity in sites of primary breast cancer using the investigational radiotracer [18F]ISO-1.

DETAILED DESCRIPTION:
This study will evaluate the feasibility of using [18F]ISO-1 PET/CT to image sigma-2 receptor binding in primary breast tumors and continue to evaluate the safety of the tracer in this patient population. [18F]ISO-1 uptake measures will be correlated with qualitative immunohistochemical staining for cell proliferation (Ki67). This is an observational study in that [18F]ISO-1 PET/CT will not be used to direct treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age
2. Known or suspected breast cancer with at least one breast lesion that is 1 cm or greater in size by standard imaging (e.g. mammography, ultrasound or breast MRI)
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures

Exclusion Criteria:

1. Females who are pregnant at the time of screening will not be eligible for this study, urine or serum pregnancy test will be performed in women of child-bearing potential at the time of screening.
2. Inability to tolerate imaging procedure in the opinion of an investigator or treating physician
3. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
4. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Correlate [18F]ISO-1 uptake with pathologic assays measuring cellular proliferation rates (e.g. Ki-67) | 6 years
  Correlate [18F]ISO-1 uptake with pathologic assays measuring cellular proliferation rates (e.g. Ki-67)

SECONDARY OUTCOMES:
Evaluate the feasibility of using [18F]ISO-1 to image sigma-2 receptor binding in breast cancer | 6 years
  Evaluate the feasibility of using [18F]ISO-1 to image sigma-2 receptor binding in breast cancer
Evaluate the safety of [18F]ISO-1 | 6 years
  Evaluate the safety of [18F]ISO-1
Correlate [18F]ISO-1 uptake with Autoradiography | 6 years
  Correlate [18F]ISO-1 uptake with Autoradiography
Correlate [18F]ISO-1 uptake a with multi-gene expression assay, validated to predict recurrence | 6 years
  Correlate [18F]ISO-1 uptake a with multi-gene expression assay, validated to predict recurrence
Correlate [18F]ISO-1 uptake with outcomes (e.g. time to recurrence, progression free survival and overall survival) | 6 years
  Correlate [18F]ISO-1 uptake with outcomes (e.g. time to recurrence, progression free survival and overall survival)
Test the association of [18F]ISO-1 uptake with phenotypic breast cancer subtypes (e.g. HER2+, TN, ER/PR+, etc.) | 6 years
  Test the association of [18F]ISO-1 uptake with phenotypic breast cancer subtypes (e.g. HER2+, TN, ER/PR+, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McDonald, MD, PhD, Principal Investigator — University of Pennsylvania; David Mankoff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] McDonald ES, Doot RK, Young AJ, Schubert EK, Tchou J, Pryma DA, Farwell MD, Nayak A, Ziober A, Feldman MD, DeMichele A, Clark AS, Shah PD, Lee H, Carlin SD, Mach RH, Mankoff DA. Breast Cancer 18F-ISO-1 Uptake as a Marker of Proliferation Status. J Nucl Med. 2020 May;61(5):665-670. doi: 10.2967/jnumed.119.232363. Epub 2019 Dec 13. PMID 31836680